CLINICAL TRIAL: NCT01744483
Title: Pilot Trial of Tubes to Prevent Ventilator-Associated Pneumonia (PreVent)
Brief Title: Endotracheal Tubes for Prevention of Ventilator-associated Pneumonia
Acronym: PreVent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Miriam Treggiari, Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 42230; 5R34HL105581-02 (NIH)
Record Dates: First submitted 2012-11-29; First posted 2012-12-06 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Ventilator-acquired Pneumonia
Keywords: pneumonia; endotracheal intubation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PVC ETT (Active Comparator): Polyvinylchloride cuff endotracheal tube
  Interventions: Device: PVC ETT
- PUC ETT (Experimental): Polyurethane cuff endotracheal tube
  Interventions: Device: PUC ETT
- PUC-CASS ETT (Experimental): Polyurethane cuff with continuous aspiration of subglottic secretions endotracheal tube
  Interventions: Device: PUC-CASS ETT

INTERVENTIONS:
Device: PVC ETT — Placement of a PVC-cuffed ETT in the setting of emergent intubation.
  Other Names: Mallinckrodt Hi-Lo Oral/Nasal ETT Cuffed. Murphy Eye.
  Arms: PVC ETT
Device: PUC ETT — Placement of a PUC-cuffed ETT in the setting of emergent intubation.
  Other Names: Mallinckrodt Seal Guard, oral/nasal ETT.
  Arms: PUC ETT
Device: PUC-CASS ETT — Placement of a PUC-cuffed in the setting of emergent intubation, followed by continuous aspiration of subglottic secretions for the duration of mechanical ventilation.
  Other Names: Mallincrodt Evac Oral ETT, Seal Guard, Murphy Eye
  Arms: PUC-CASS ETT

SUMMARY:
Researchers are looking at three different types of breathing tubes to see if any of them are better at preventing pneumonia than the others. Two of the tubes have design features to prevent leakage of fluids from the mouth and throat into the lungs. This is importance, since leakage of small amounts of fluid into the lungs may lead to pneumonia. The third tube is the standard tube used at most hospitals.

The hypothesis is that the use of a breathing tube that reduces fluid leakage into the lungs will reduce the risk of developing pneumonia, compared to the standard tube. The study will also look at the safety of the modified breathing tubes, compared to the standard tube.

This study is a small, "pilot" study that will determine if it is possible to perform a larger study that will provide more certain results.

DETAILED DESCRIPTION:
The objective of this pilot study is provide data for planning and to establish the feasibility of performing a large, randomized, comparative effectiveness trial of two specially designed airway tubes (endotracheal tubes; ETTs) for the prevention of ventilator-associated pneumonia (VAP). Modification of the material and design of the ETT cuff that is positioned in the trachea, and/or continuous aspiration of subglottic secretions through an extra port positioned between the tube cuff and the vocal chords may prevent leakage of contaminated secretions around the cuff and thereby reduce the risk of VAP. The investigators are planning a phase III, randomized, controlled trial comparing the effectiveness of a polyurethane-cuffed endotracheal tube (PUC-ETT), a polyurethane-cuffed tube that also allows continuous aspiration of subglottic secretions (PUC-CASS-ETT), and a conventional, polyvinylchloride-cuffed endotracheal tube (PVC-ETT) in mechanically ventilated patients with respiratory failure. Prior to initiating the Phase III trial, a smaller pilot study is necessary in order to establish feasibility and to gather data on endpoints in order to establish enrollment rates and project sample size for the definitive trial. For the purposes of planning, a surrogate for VAP, bacterial colonization of the trachea will be assessed from daily quantitative cultures to allow estimation of effect size for the two study devices. VAP will be diagnosed using objective criteria, based on cultures from bronchoalveolar lavage. The safety profile of the tubes will be evaluated using a multi-faceted approach, including short-term objective measures of laryngeal dysfunction and long-term subjective and objective assessment of upper airway problems via phone interview post-hospital discharge, and recording of device-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Emergency intubation with a study device either in the field by Medic One, (the Seattle Fire Department program that provides basic and advanced life support services to the city) or at HMC;
3. Absence of out-of-hospital cardiac arrest;
4. Absence of major burns, penetrating trauma or absence any major trauma with systolic blood pressure < 90 mmHg at the time of tracheal intubation.

Exclusion Criteria:

1. Use of a non-study designated intubation device (such as nasal intubation, tracheostomy, intubation in the operating room, intubation outside the study network such as occurring in an outside hospital or by other emergency response providers);
2. Patients with permanent tracheostomy;
3. Federally protected populations: Children (age <18 years), pregnant women, and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Treggiari, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Deem S, Yanez D, Sissons-Ross L, Broeckel JA, Daniel S, Treggiari M. Randomized Pilot Trial of Two Modified Endotracheal Tubes To Prevent Ventilator-associated Pneumonia. Ann Am Thorac Soc. 2016 Jan;13(1):72-80. doi: 10.1513/AnnalsATS.201506-346OC. PMID 26523433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing emergency tracheal intubation. EMS routed Harborview Medical Center (HMC) or patients who required emergent tracheal intubation while in HMC.
Period: Overall Study
Arm/Group | PVC ETT | PUC ETT | PUC-CASS ETT
Started | 44 | 35 | 38
Completed | 15 | 13 | 10
Not Completed | 29 | 22 | 28
Not completed — Death | 9 | 4 | 11
Not completed — Lost to Follow-up | 8 | 9 | 11
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 6 | 2
Not completed — No ICU Admit | 5 | 1 | 2
Not completed — Routed to OSH | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Figures do not include inadvertent enrollments (IRB excluded, Not admitted to ICU or Routed to OSH)
Groups:
- Total: Total of all reporting groups
Arm/Group | PVC ETT | PUC ETT | PUC-CASS ETT | Total
Number analyzed (Participants) | 36 | 32 | 34 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 25 | 28 | 75
  >=65 years | 14 | 7 | 6 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 10 | 30
  Male | 27 | 21 | 24 | 72
Region of Enrollment [Number; unit: participants]
  United States | 36 | 32 | 34 | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Tracheal Bacterial Colonization
Description: The percentage of patients with quantitative culture growth from tracheal aspirate specimens of >1,000,000 CFU between Day 2 and Day 4 of tracheal intubation/mechanical ventilation. Percentage of patients will be compared between the three study arms.
Time Frame: Tracheal colonization by Day 4 or extubation
Measure: Number; unit: percentage of tracheal colonization
Arm/Group | PVC ETT | PUC ETT | PUC-CASS ETT
Number analyzed (Participants) | 33 | 29 | 34
percentage of tracheal colonization | 8 | 7 | 9

ADVERSE EVENTS:
Time Frame: Up to 2 months after extubation
Description: Death or prolonged hospitalization related to ETT model
Arm/Group | PVC ETT | PUC ETT | PUC-CASS ETT
Serious Adverse Events (participants affected / at risk) | 9/36 | 5/32 | 9/34
Other Adverse Events (participants affected / at risk) | 1/36 | 1/32 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PVC ETT (N=36) | PUC ETT (N=32) | PUC-CASS ETT (N=34)
Death from any cause (Cardiac disorders) | 9 (9) | 5 (5) | 9 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PVC ETT (N=36) | PUC ETT (N=32) | PUC-CASS ETT (N=34)
Up to 2 months after extubation airway complications (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes